CLINICAL TRIAL: NCT01788553
Title: An Observational Study of Remission in Patients Treated for Generalized Anxiety Disorder in Primary and Specialized Care in Belgium.
Brief Title: Study Of Remission In Patients Treated For Generalized Anxiety Disorder
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0600B-102246; B2411129 (Other: Pfizer)
Record Dates: First submitted 2009-07-06; First posted 2013-02-11 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Anxiety Disorders
Keywords: remission; generalized anxiety disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with generalized anxiety disorder
  Interventions: Other: remission prevalence of generalized anxiety disorder

INTERVENTIONS:
Other: remission prevalence of generalized anxiety disorder

SUMMARY:
The aim of the study is to assess the remission rates in patients treated for generalized anxiety disorder in primary and specialized care. Factors that may influence remission such as disease history and severity of the anxiety disorder, the type of treatment, the presence of co-morbid depression or anxiety disorder as well as socio-demographic factors will also be evaluated. The study will also assess patient functioning and compare functioning in patients who do and do not achieve remission.

DETAILED DESCRIPTION:
The aim of the study is to assess the remission rates in patients treated for generalized anxiety disorder in primary and specialized care. Factors that may influence remission such as disease history and severity of the anxiety disorder, the type of treatment, the presence of co-morbid depression or anxiety disorder as well as socio-demographic factors will also be evaluated. The study will also assess patient functioning and compare functioning in patients who do and do not achieve remission.

The objectives of the study are:

Primary: To determine the prevalence of remission in patients treated for generalized anxiety disorder in primary care and specialized care. Secondary: To determine patient functioning and work loss days and compare these in patients who do or do not achieve remission. To determine the effect of disease factors on remission rate such as disease history, duration, severity, co-morbidity with depression or other anxiety disorders. To determine the effect of treatment factors on remission rate such as setting, type of treatment, duration and adherence. To determine the effect of socio-demographic factors on remission rate such as gender, age, region (language), marital status, educational level and employment status.

This will be a cross-sectional observational study looking at the point prevalence of remission in treated patients with generalized anxiety disorder in general practice and specialized care in Belgium. General practitioners and psychiatrists will assess remission rates in patients treated for generalized anxiety disorder during 1 routine visit of these patients.

The participating physicians will have 3 months to evaluate remission at a routine visit in 5 to 10 patients that have been treated for generalized anxiety disorder since at least 3 months

ELIGIBILITY:
Inclusion criteria:

To be eligible the patient must meet all of the following:

1. Being treated for generalized anxiety disorder for approximately 3 months and not more than 12 months
2. Be at least 18 years of age;
3. Written informed consent
4. Out-patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with generalized anxiety disorder in primary and specialized care in Belgium.
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2006-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
remission of generalized anxiety disorder | 5 months

SECONDARY OUTCOMES:
determine the effect of disease and treatment factors on remission rates | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Pfizer Inc., Brussels, Belgium